CLINICAL TRIAL: NCT05725629
Title: The Study Was Conducted According to the Guidelines of the Declaration of Helsinki, and Approved by the Institutional Review Board (IRB Number: 201900999B0) of the Chang Gung Medical Foundation.
Brief Title: Discussion on the Association Model of Traditional Chinese Medi-cine Body Constitution and Female Infertility
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Pei-Hung Liao, Associate professor, National Taipei University of Nursing and Health Sciences
Other Study IDs: 201900999B0
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Association Model; Chinese Medicine Physique Types; Health Care Base on Traditional Chinese Medicine; Women Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Abstract Background: Infertility may cause physiological and psychological distress. The Health Promotion Administration in Taiwan has listed infertility improvement under the "Reproductive health and prevention section" in the Whole Person Wellness policy.

Methods: This study was based on an exploratory research design. It used artificial intelligence algorithms such as logistic regression and association rules, and constructed the association model between the physique literature of traditional Chinese medicine and common demographic variables.

Results: The participants showed three types of constitutions in traditional Chinese medicine, namely Yin deficiency, Yang deficiency, and phlegm stasis. Infertile women who prefer to eat heavy or sour-tasting foods were 2.8 times more likely to have ovarian factors than those who do not like to eat those foods.

Conclusions: Based on the correction between physique type and the demographic variables of infertile women, care based on traditional Chinese medicine should be pro-vided to improve the body constitutions of infertile women.

DETAILED DESCRIPTION:
Abstract Background: Infertility may cause physiological and psychological distress. The Health Promotion Administration in Taiwan has listed infertility improvement under the "Reproductive health and prevention section" in the Whole Person Wellness policy.

Methods: This study was based on an exploratory research design. It used artificial intelligence algorithms such as logistic regression and association rules, and constructed the association model between the physique literature of traditional Chinese medicine and common demographic variables.

Results: The participants showed three types of constitutions in traditional Chinese medicine, namely Yin deficiency, Yang deficiency, and phlegm stasis. Infertile women who prefer to eat heavy or sour-tasting foods were 2.8 times more likely to have ovarian factors than those who do not like to eat those foods.

Conclusions: Based on the correction between physique type and the demographic variables of infertile women, care based on traditional Chinese medicine should be pro-vided to improve the body constitutions of infertile women.

ELIGIBILITY:
Inclusion Criteria:

* Female

Exclusion Criteria:

* male

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The purpose of this study was to explore the physique of infertile women in Taiwan and their association with TCM body constitution.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
understand the physiques of infertile women through TCM. | 2019~2023
  TCM physiques are significantly related to the causes of infertility, but infertility women can change their daily habits to change their physiques and maintain their health. Therefore, it is particularly important to improve the understanding of basic TCM nursery care for infertile women

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided